CLINICAL TRIAL: NCT01895452
Title: A Phase 3, Multicenter Extension of Study ALK9072-003EXT to Assess the Long-term Safety and Durability of Effect of ALKS 9072 in Subjects With Stable Schizophrenia
Brief Title: An Extension of a Long-term Safety Study of ALKS 9072 (Also Known as ALKS 9070)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK9072-003EXT2
Record Dates: First submitted 2013-07-05; First posted 2013-07-10 (Estimated); Results first posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALKS 9072, Low Dose (Experimental)
  Interventions: Drug: ALKS 9072, Low Dose
- ALKS 9072, High Dose (Experimental)
  Interventions: Drug: ALKS 9072, High Dose

INTERVENTIONS:
Drug: ALKS 9072, Low Dose — Intramuscular injection, given monthly
  Arms: ALKS 9072, Low Dose
Drug: ALKS 9072, High Dose — Intramuscular injection, given monthly
  Arms: ALKS 9072, High Dose

SUMMARY:
This is an extension of a previous study (ALK9072-003EXT). The purpose of this study is to continue to evaluate the long-term safety and durability of effect of ALKS 9072 in subjects with stable schizophrenia, and to allow subjects who are doing well on ALKS 9072 to continue treatment.

ELIGIBILITY:
Inclusion Criteria:

* Completed the treatment period of Study ALK9072-003EXT
* Continues to require chronic treatment with an antipsychotic medication
* Continues to reside in a stable living situation
* Continues to have an identified reliable informant

Exclusion Criteria:

* Abnormal clinical laboratory value, vital sign, or electrocardiogram (ECG) finding during participation in Study ALK9072-003EXT that was clinically relevant and related to study drug
* Missed more than 1 scheduled study visit during participation in the preceding Study ALK9072-003EXT
* Has a significant or unstable medical condition that would preclude safe completion of the current study
* Subject is pregnant or breastfeeding
* Subject expects to be incarcerated, or has pending legal action which may impact compliance with study participation or procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Risinger, MD, Study Director — Alkermes, Inc.
Locations (54):
- United States (14):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, Oakland, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, Washington D.C., District of Columbia
  - Alkermes Investigational Site, Fort Lauderdale, Florida
  - Alkermes Investigational Site, Leesburg, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Hoffman Estates, Illinois
  - Alkermes Investigational Site, Shreveport, Louisiana
  - Alkermes Investigational Site, Oklahoma City, Oklahoma
  - Alkermes Investigational Site, Dallas, Texas
- Bulgaria (8):
  - Alkermes Investigational Site, Burgas
  - Alkermes Investigational Site, Novi Iskar
  - Alkermes Investigational Site, Pazardzhik
  - Alkermes Investigational Site, Plovdiv
  - Alkermes Investigational Site, Sofia
  - Alkermes Investigational Site, Targovishte
  - Alkermes Investigational Site, Veliko Tarnovo
  - Alkermes Investigational Site, Vratsa
- Malaysia (4):
  - Alkermes Investigational Site, Cheras
  - Alkermes Investigational Site, Johor Bahru
  - Alkermes Investigational Site, Kuala Lampur
  - Alkermes Investigational Site, Kuching
- Philippines (5):
  - Alkermes Investigational Site, Mariveles, Bataan
  - Alkermes Investigational Site, Cebu City
  - Alkermes Investigational Site, Iloilo City
  - Alkermes Investigational Site, Mandaluyong
  - Alkermes Investigational Site, Manila
- Romania (3):
  - Alkermes Investigational Site, Bucharest
  - Alkermes Investigational Site, Oradea
  - Alkermes Investigational Site, Târgu Mureş
- Russia (10):
  - Alkermes Investigational Site, Roshchino, Vyborgskiy
  - Alkermes Investigational Site, Lipetsk
  - Alkermes Investigational Site, Moscow
  - Alkermes Investigational Site, Rostov-on-Don
  - Alkermes Investigational Site, Saint Petersburg
  - Roshchino township, Samara
  - Roshchino township, Saratov
  - Alkermes Investigational Site, Stavropol
  - Alkermes Investigational Site, Talagi
  - Alkermes Investigational Site, Yaroslavl
- Alkermes Investigational Site, Jeollanam-do, South Korea
- Ukraine (9):
  - Alkermes Investigational Site, Chernihiv
  - Alkermes Investigational Site, Donetsk
  - Alkermes Investigational Site, Kharkiv
  - Alkermes Investigational Site, Kherson
  - Alkermes Investigational Site, Kyiv
  - Alkermes Investigational Site, Lviv
  - Alkermes Investigational Site, Poltava
  - Alkermes Investigational Site, Ternopil
  - Roshchino township, Vinnytsia

REFERENCES:
- [Derived] McEvoy JP, Weiden PJ, Lysaker PH, Sun X, O'Sullivan AK. Long-term effect of aripiprazole lauroxil on health-related quality of life in patients with schizophrenia. BMC Psychiatry. 2021 Mar 24;21(1):164. doi: 10.1186/s12888-021-03124-2. PMID 33761928
- [Derived] Lauriello J, Claxton A, Du Y, Weiden PJ. Beyond 52-Week Long-Term Safety: Long-Term Outcomes of Aripiprazole Lauroxil for Patients With Schizophrenia Continuing in an Extension Study. J Clin Psychiatry. 2020 Aug 18;81(5):19m12835. doi: 10.4088/JCP.19m12835. PMID 32841554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who successfully completed the treatment period in Study ALK9072-003EXT and continued to meet eligibility criteria were eligible to enroll in this extension study.
Groups:
- ALKS 9072, Low: ALKS 9072, Low : IM injection, given monthly
- ALKS 9072, High: ALKS 9072, High: IM injection, given monthly
Period: Overall Study
Arm/Group | ALKS 9072, Low | ALKS 9072, High
Started | 65 | 226
Completed | 61 | 198
Not Completed | 4 | 28
Not completed — Adverse Event | 1 | 4
Not completed — Lost to Follow-up | 1 | 5
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 2 | 14
Not completed — Underlying disease | 0 | 3
Not completed — Noncompliance with study drug | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population includes all subjects who received at least 1 dose of ALKS 9072 in the current study.
Groups:
- Total: Total of all reporting groups
Arm/Group | ALKS 9072, Low | ALKS 9072, High | Total
Number analyzed (Participants) | 65 | 226 | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (11.02) | 40.1 (11.59) | 39.6 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 107 | 135
  Male | 37 | 119 | 156
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 49 | 65
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 19 | 21
  White | 47 | 157 | 204
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 0 | 5 | 5
  Romania | 2 | 1 | 3
  United States | 4 | 32 | 36
  Philippines | 15 | 27 | 42
  Ukraine | 15 | 64 | 79
  Malaysia | 1 | 17 | 18
  Bulgaria | 13 | 32 | 45
  Russia | 15 | 48 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: This measure includes all incidences, including those that occurred >5%.
Time Frame: Up to 12 months
Population: Safety population includes all subjects who received at least 1 dose of ALKS 9072 in the current study.
Measure: Count of Participants; unit: Participants
Arm/Group | ALKS 9072, Low | ALKS 9072, High
Number analyzed (Participants) | 65 | 226
Participants | 21 | 94

2. Secondary Outcome: Change in Baseline of Positive and Negative Syndrome Scale (PANSS) Total Score Over Time
Description: This scale consists of symptom constructs (7 positive, 7 negative, 16 general psychopathology), each to be rated on a 7-point Likert-type scale of severity with 1 being absent to 7 being extreme. Minimum scores (best outcome) equals 30 (total scale); maximum scores (worst outcome) equals 210 (total scale). Change is calculated between the baseline visit and the subject's last visit in the treatment period.
Time Frame: Up to 12 months
Population: The full analysis set consisted of all subjects who received at least 1 dose of ALKS 9072 and had at least 1 postbaseline assessment of PANSS total score after administration of ALKS 9072.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALKS 9072, Low | ALKS 9072, High
Number analyzed (Participants) | 65 | 221
units on a scale | -0.7 (6.73) | -0.9 (6.07)

3. Secondary Outcome: Mean Change From Baseline to Endpoint in Clinical Global Impression - Severity (CGI-S) Over Time
Description: The CGI-S is a 7-point scale that requires the clinician to assess how mentally ill the patient is in a specific point in time. Results indicate participants evaluated at one of the following categories: "1: normal, not at all ill"; "2: borderline mentally ill"; "3: mildly ill"; "4: moderately ill"; "5: markedly ill"; "6: severely ill"; and "7: among the most extremely ill patients". Results indicate a change in CGI-S score from baseline to Day 365 based on the observed data. Change is calculated between the baseline visit and the subject's last visit in the treatment period.
Time Frame: Up to 12 months
Population: The full analysis set consists of all subjects who received at least 1 dost of ALKS 9072 and had at least 1 postbaseline assessment of PANSS score after administration of ALKS 9072.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALKS 9072, Low | ALKS 9072, High
Number analyzed (Participants) | 65 | 221
units on a scale | -0.1 (0.48) | -0.1 (0.52)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at every study visit for up to 35 months.
Arm/Group | ALKS 9072, Low | ALKS 9072, High
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/226
Serious Adverse Events (participants affected / at risk) | 0/65 | 4/226
Other Adverse Events (participants affected / at risk) | 11/65 | 26/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALKS 9072, Low (N=65) | ALKS 9072, High (N=226)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1) — worsening/exacerbation of schizophrenia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALKS 9072, Low (N=65) | ALKS 9072, High (N=226)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 7 (8)
Toothache (Gastrointestinal disorders) | 4 (4) | 3 (4)
Nasopharyngitis (Infections and infestations) | 4 (4) | 9 (11)
Insomnia (Psychiatric disorders) | 2 (4) | 16 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.